## Effect of Semaglutide on the Psoriatic Lesion in Patients

## With Type 2 Diabetes Mellitus

Date 08.may 2023

## Statistical analysis

Descriptive statistics will be presented via mean and standard deviation (SD) for continuous variables and percentages for categorical variables. To compare the mean value, i.e. median for continuous parameters between group 1 and group 2, the t-test for two independent samples, i.e. the Wilcoxon Mann–Whitney test for two independent groups will be used. Spearman's correlation analysis will be used to determine the correlation between parameters. Chi-square test will be used for categorical parameters. To determine the significance of the correlation, binary logistic regression will be used in order to find the influence of the independent variable (predictor-factor) on the dependent variable (presence of arthritis; presence of comorbidities; severity of the disease). Statistical testing of hypotheses was done with two-sided statistical tests with a statistical significance level of 5%. All results will be presented tabularly and graphically.